CLINICAL TRIAL: NCT06107660
Title: Utility of Exparel Based Erector Spinae Plane Block for Elective 1 and 2 Level Posterior-based Lumbar Fusion: A Randomized Control Trial
Brief Title: Utility of Exparel Based ESP Blocks in Elective Posterior Spine Fusion
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hartford Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HHC-2023-0204
Record Dates: First submitted 2023-10-18; First posted 2023-10-30 (Actual); Last update posted 2023-10-30 (Actual); Status verified 2023-10

CONDITIONS: Spine Fusion; Anesthesia, Local
Keywords: Erector Spinae Block; Lumbar Spine; bupivacaine; Exparel
MeSH Terms: interventions — Bupivacaine

STUDY DESIGN:
Intervention Model Description: Enrolled participants will be randomized to receive either a mixture of liposomal bupivacaine/ bupivacaine or standard bupivacaine with adjuncts for their ESPB.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The patient, orthopedic surgeon (investigator or care provider), and outcome assessor performing data analysis will be blinded to this study. The regional anesthesia block is performed prior to surgical incision without the surgeon present, and thus the surgeon will be blinded to which formulation was provided. The patient will be informed that they are receiving a block but will not be informed until data collection is complete at the 3 month mark as to which group they were part of.
  Non-blinded Parties: Due to differences in the physical appearance it is impossible to blind the anesthesia team (attending and fellow) performing the block, as the standard block is clear while the Exparel formulation is milky. However, after the regional block has been performed the regional team will have no further contact with the patient as per standard practice, and thus maintaining a separation between those blinded and not.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Study Group (Experimental): Patients in the study Group will receive 20ml 1.3% Liposomal bupivacaine (Exparel®) dose of 266mg with 40 ml of 0.25% bupivacaine.
  The local anesthetic solution will be administered bilaterally in the plane between the lumber transverse process and the erector spinae muscles to block the dorsal and ventral rami of the spinal nerves under ultrasound guidance using a standard block needled. A total of 60 ml solution will be injected -30 ml on each side of the spinal column.
  Interventions: Drug: Liposomal bupivacaine
- Control Group (Active Comparator): Patients in the control group will receive 60ml of 0.25% bupivacaine with 5 mg preservative free dexamethasone and 150 mcg Epinephrine (in a 1:400,000 dilution).
  The local anesthetic solution will be administered bilaterally in the plane between the lumber transverse process and the erector spinae muscles to block the dorsal and ventral rami of the spinal nerves under ultrasound guidance using a standard block needled. A total of 60 ml solution will be injected -30 ml on each side of the spinal column.
  Interventions: Drug: Bupivacaine

INTERVENTIONS:
Drug: Liposomal bupivacaine — Patients will receive either liposomal bupivacaine as part of the ESPB .
  Other Names: Exparel
  Arms: Study Group
Drug: Bupivacaine — This is the control group comparator as this is standard of care at the investigator's institution.
  Arms: Control Group

SUMMARY:
The goal of this clinical trial is to compare two different medications used to reduce pain during lower back fusion surgery. The main questions this study aims to answer are:

1. Can liposomal bupivacaine, when included in a regional anesthesia technique called the Erector Spinae Plane block (ESPB), reduce opioid use post-operatively compared to the standard medication typically used in an ESPB (bupivacaine with stabilizing agents)?
2. Do patients report lower pain and better satisfaction with their surgery when they receive liposomal bupivacaine in the ESPB compared to those that receive the standard medication?

Participants will be randomized to into two groups one that receives liposomal bupivacaine and one group that receives bupivacaine with stabilizing agents. Other than the randomization all patients will follow current standard of care at our hospital, and will not be asked to complete any additional study forms in addition to forms currently asked of all patients as per standard of care.

DETAILED DESCRIPTION:
The purpose of this study is to improve pain management for patients having spine fusion surgery. This aim will be achieved by evaluating how well liposomal bupivacaine (LB), an FDA approved numbing medication that can provide pain relief for up to 72 hours after surgery, works when used as a single dose in a regional block known as Erector Spinae Plane block (ESPB). ESPB is a regional anesthesia technique used to control pain after surgery by injecting numbing medication around the patient's back bones on both sides. The study will compare how well LB in ESPB works compared to the standard practice procedure, which involves administering the traditional numbing medication (bupivacaine) through the ESPB. These two medications will be evaluated in reducing postoperative opioid medication need to control postoperative pain, as the primary goal. This study seeks to understand whether an ESP block either with bupivacaine and stabilizing agents or using liposomal bupivacaine, reduces the total amount of opioid medication used postoperatively, reduces pain scores, and leads to better patient reported outcome scores, patient satisfaction, and reduced recovery time in the PACU. Should the investigator find that liposomal bupivacaine is not superior to bupivacaine with stabilizing agents, this information would prove useful in regards to analgesic options for this patient population and could lead to a substantial cost savings.

ELIGIBILITY:
Inclusion Criteria:

* Lumbar pathology requiring a single or two level elective posterior based (i.e. posterior or transforaminal approach) spine fusion with or without an interbody device.
* Surgical approach through either a midline or paramedian incision
* Primary fusion surgery, previous decompression surgery is acceptable
* American Society of Anesthesiologists (ASA) score of 1,2,or 3.

Exclusion Criteria:

* Patients currently on narcotic pain medication for pain management
* Patients with a history of illicit drug use
* Patients with neuromuscular disorders or neurological deficits (i.e. post polio or myasthenia gravis)
* Patients confined to a wheelchair for over 6 months
* Patients with fibromyalgia or other chronic pain disorder
* Patient with contraindications for use of the ESP block (i.e. local skin infection over the area of needle entry, or anaphylactic reaction to bupivacaine)
* Non-invasive surgical approaches
* Repeat or revision surgery
* Non-posterior spine surgical approaches (i.e. lateral, oblique, anterior, anterior and posterior approaches)
* Staged procedures
* Adjacent segment surgery
* Patients with a weight less than 40kg to avoid local anesthetic systematic toxicity.

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-12 (Estimated); Primary Completion 2025-06 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Opioid Use | 72 hours (standard inpatient stay)
  Opioid Use in patient stay measured in morphine milligram equivalents

SECONDARY OUTCOMES:
Pain Report at Rest-Immediate postop | Asked immediately after surgery while patient is recovering in the post-anesthesia care unit (PACU).
  Pain as measured using Numeric Pain Scale (NPS) while patient is at rest immediate postoperative. The minimum value on the NPS is 0 indicating no pain (best outcome) and 10 indicates severe pain (worst outcome)
Pain Report with activity-Immediate postop | Patient is asked their pain level once they have been moved to their hospital room from the PACU. Typically this occurs within 5 hours of surgery.
  Pain as measured using Numeric Pain Scale (NPS) while patient is active immediate postoperative. The minimum value on the NPS is 0 indicating no pain (best outcome) and 10 indicates severe pain (worst outcome)
Pain Report at Rest-Post op day 1 | 24 hours post-op
  Pain as measured using Numeric Pain Scale (NPS) while patient is at rest 24 hours after surgery. The minimum value on the NPS is 0 indicating no pain (best outcome) and 10 indicates severe pain (worst outcome).
Pain Report with activity-Post op day 1 | 24 hours post-op
  Pain as measured using Numeric Pain Scale (NPS) with activity 24 hours after surgery. The minimum value on the NPS is 0 indicating no pain (best outcome) and 10 indicates severe pain (worst outcome).
Pain Report at rest-at discharge | 72 hours post-op
  Pain as measured using Numeric Pain Scale (NPS) while patient is at rest at discharge. The minimum value on the NPS is 0 indicating no pain (best outcome) and 10 indicates severe pain (worst outcome).
Pain Report with activity-at discharge | 72 hours post-op
  Pain as measured using Numeric Pain Scale (NPS) with activity at discharge. The minimum value on the NPS is 0 indicating no pain (best outcome) and 10 indicates severe pain (worst outcome).
PACU recovery time | <5 hours post op
  Time from entry into PACU to time patient is listed as recovered
Patient Statisfcation | 10-14 days post-op
  Based on Press Ganey Patient Satisfaction Survey. The minimum score is 0 (very poor) while the maximum score is 100 (very good).
Patient reported outcomes score | 3 months post-op
  Oswestry Disability Index (ODI) score. The minimum ODI score is 0 and represents minimal disability, while the maximum score of 100 represents the worst outcome - bed-bound significant disability.

CONTACTS AND LOCATIONS:
Overall Officials: Heeren Makanji, MD, Principal Investigator — Hartford HealthCare

IPD SHARING:
Plan to Share IPD: No
No individual participant data will be shared as part of this study.

REFERENCES:
- [Background] Makanji HS, Solomito MJ, Maffeo-Mitchell C, Esmende S, Finkel K. Utility of Erector Spinae Plane Blocks for Postoperative Pain Management and Opioid Reduction Following Lumbar Fusions. Clin Spine Surg. 2023 May 1;36(4):E131-E134. doi: 10.1097/BSD.0000000000001387. Epub 2022 Sep 13. PMID 36097343